CLINICAL TRIAL: NCT00095303
Title: Brief Strategic Family Therapy for Adolescent Drug Abusers
Acronym: BSFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Oregon Research Institute (Other)
Responsible Party: Principal Investigator, Jose Szapocznik, Chair, Department of Epidemiology and Public Health, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20090698; U10DA013720 (NIH); 5RC2DA028864 (NIH)
Record Dates: First submitted 2004-11-02; First posted 2004-11-03 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Substance Abuse
Keywords: BSFT; Family Therapy; Adolescents; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief Strategic Family Therapy (BSFT) (Experimental): BSFT is a family therapy approach that consists of 12 to 16 sessions (each 1 to 1.5 hours long) over a 4-month period during the Main Study, and up to 8 "booster" sessions. Interventions are delivered to adolescents and relevant family members in non-restrictive community settings (e.g., clinics, homes, school).
  Interventions: Behavioral: Brief Strategic Family Therapy (BSFT)
- Treatment as Usual (TAU) (Active Comparator): TAU varies depending on site, however each will offer services that include at least 1 therapy session (individual or group therapy) per week during the Main Study, as well as participation in ancillary services (e.g., case management, self help groups, etc.) over a four month period.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Brief Strategic Family Therapy (BSFT) — BSFT is a family therapy approach that consists of 12 to 16 sessions (each 1 to 1.5 hours long) over a 4-month period during the Main Study, and up to 8 "booster" sessions. Interventions are delivered to adolescents and relevant family members in non-restrictive community settings (e.g., clinics, homes, school).
  Other Names: BSFT
  Arms: Brief Strategic Family Therapy (BSFT)
Behavioral: Treatment as Usual — TAU varies depending on site, however each will offer services that include at least 1 therapy session (individual or group therapy) per week during the Main Study, as well as participation in ancillary services (e.g., case management, self help groups, etc.) over a four month period.
  Other Names: TAU
  Arms: Treatment as Usual (TAU)

SUMMARY:
The purpose of this study is to compare Brief Strategic Family Therapy (BSFT) for Adolescent Drug Abusers to treatment as usual (TAU).

An additional follow up assessment, funded by an American Recovery & Reinvestment Act (ARRA) grant, was completed 5 years post randomization in order to examine the long term effects of outpatient treatments for illicit drug using adolescents.

DETAILED DESCRIPTION:
Adolescent drug abuse continues to be one of the most pressing public health issues in the United States-our nation's teenagers continue to use illicit drugs at a worrisome rate. Broad reviews of the treatment outcome literature indicate that family interventions in general, and Brief Strategic Family Therapy (BSFT) in particular, are effective with drug using youth. This study is designed to compare BSFT to treatment as usual (TAU). The researchers believe that BSFT will be much more effective than TAU in reducing adolescent drug use. They will also examine which of these treatment approaches does a better job of engaging adolescents and family members in treatment, decreasing problem behaviors, decreasing sexually risky behaviors, increasing pro-social activities (e.g., school, work), and improving the functioning of the family.

With the addition of the extended follow up, we have the opportunity to examine the sustainability of study outcomes into early adulthood, filling a gap in the treatment research literature about the long-term effects of adolescent substance abuse treatment. The follow up study examined the long term effectiveness of BSFT compared to TAU in the rates of substance use, number of arrests and externalizing behaviors, in youth who received study treatments at the time when they were adolescents.

ELIGIBILITY:
Main Study:

Inclusion Criteria:

* adolescents ages 12 to 17
* used any illicit drugs (other than alcohol and tobacco) in the 30-day period
* live with or intend to live with a formal or informal family

Exclusion Criteria:

* suicidal or homicidal ideation.

Follow Up Study:

Inclusion Criteria:

* youth must have signed consent during the main study to be approached for future research
* currently 18 years old or older

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2004-08; Primary Completion 2008-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Szapocznik, Ph.D., Principal Investigator — University of Miami
Locations (8):
- United States (7):
  - La Frontera Center, Tucson, Arizona
  - Tarzana Treatment Center, Tarzana, California
  - Arapahoe House, Thornton, Colorado
  - Gateway Community Services, Jacksonville, Florida
  - The Villiage, Miami, Florida
  - Daymark, Concord, North Carolina
  - The Crossroads Center, Cincinnati, Ohio
- Centro de Salud Mental de la Comunidad de Bayamsn, Bayamón, Puerto Rico

REFERENCES:
- [Background] Horigian VE, Robbins MS, Dominguez R, Ucha J, Rosa CL. Principles for defining adverse events in behavioral intervention research: lessons from a family-focused adolescent drug abuse trial. Clin Trials. 2010 Feb;7(1):58-68. doi: 10.1177/1740774509356575. PMID 20156957
- [Background] Robbins MS, Alonso E, Horigian VE, Bachrach K, Burlew K, Carrion IS, Hodgkins CC, Miller M, Schindler E, VanDeMark N, Henderson C, Szapocznik J. Transporting clinical research to community settings: designing and conducting a multisite trial of brief strategic family therapy. Addict Sci Clin Pract. 2010 Dec;5(2):54-61. PMID 22002455
- [Background] Robbins MS, Feaster DJ, Horigian VE, Puccinelli MJ, Henderson C, Szapocznik J. Therapist adherence in brief strategic family therapy for adolescent drug abusers. J Consult Clin Psychol. 2011 Feb;79(1):43-53. doi: 10.1037/a0022146. PMID 21261433
- [Result] Robbins MS, Feaster DJ, Horigian VE, Rohrbaugh M, Shoham V, Bachrach K, Miller M, Burlew KA, Hodgkins C, Carrion I, Vandermark N, Schindler E, Werstlein R, Szapocznik J. Brief strategic family therapy versus treatment as usual: results of a multisite randomized trial for substance using adolescents. J Consult Clin Psychol. 2011 Dec;79(6):713-27. doi: 10.1037/a0025477. Epub 2011 Oct 3. PMID 21967492
- [Result] Weems CF, Feaster DJ, Horigian VE, Robbins MS. Parent and child agreement on anxiety disorder symptoms using the DISC predictive scales. Assessment. 2011 Jun;18(2):213-6. doi: 10.1177/1073191110389278. Epub 2010 Nov 12. PMID 21075957
- [Result] Robbins MS, Szapocznik J, Horigian VE, Feaster DJ, Puccinelli M, Jacobs P, Burlew K, Werstlein R, Bachrach K, Brigham G. Brief strategic family therapy for adolescent drug abusers: a multi-site effectiveness study. Contemp Clin Trials. 2009 May;30(3):269-78. doi: 10.1016/j.cct.2009.01.004. Epub 2009 Jan 18. PMID 19470315
- [Derived] Horigian VE, Feaster DJ, Brincks A, Robbins MS, Perez MA, Szapocznik J. The effects of Brief Strategic Family Therapy (BSFT) on parent substance use and the association between parent and adolescent substance use. Addict Behav. 2015 Mar;42:44-50. doi: 10.1016/j.addbeh.2014.10.024. Epub 2014 Nov 4. PMID 25462653
- [Derived] Horigian VE, Weems CF, Robbins MS, Feaster DJ, Ucha J, Miller M, Werstlein R. Reductions in anxiety and depression symptoms in youth receiving substance use treatment. Am J Addict. 2013 Jul-Aug;22(4):329-37. doi: 10.1111/j.1521-0391.2013.12031.x. PMID 23795871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Main Study: Adolescents who self-reported illicit drug use in the 30-days before baseline assessment or had to be referred from an institution for the treatment of drug abuse. Extended Follow Up Study: Participants from the Main Study who agreed to be contacted in the future, regardless of Main completion, were recruited to complete the assessment.
Groups:
- BSFT: Brief Strategic Family Therapy For Adolescent Drug Abusers : BSFT is a family therapy approach that consists of 12 to 16 sessions (each 1 to 1.5 hours long) over a 4-month period, and up to 8 "booster" sessions. Interventions are delivered to adolescents and relevant family members in non-restrictive community settings (e.g., clinics, homes, school).
- Treatment as Usual: Treatment as Usual : TAU varies depending on site, however each will offer services that include at least 1 therapy session per week (individual or group therapy) as well as participation in ancillary services (e.g., case management, self help groups, etc.) over a four month period.
Period: Main Study
Arm/Group | BSFT | Treatment as Usual
Started | 245 | 235
Completed | 154 | 148
Not Completed | 91 | 87
Not completed — Lost to Follow-up | 91 | 87
Period: Follow Up Study
Arm/Group | BSFT | Treatment as Usual
Started | 199 (199 (BSFT) gave permission for future contact; not a requirement to finish Main to start Follow up) | 179 (179 (TAU) gave permission for future contact; not a requirement to finish Main to start Follow up)
Completed | 140 | 121
Not Completed | 59 | 58
Not completed — Lost to Follow-up | 59 | 58

BASELINE CHARACTERISTICS:
Population: Main Study
Groups:
- BSFT: BSFT: Brief Strategic Family Therapy. 12-16 sessions, ranging from 8 to 24 as full dose Sessions include adolescents and family members
- TAU- Treatment as Usual: TAU: Treatment As Usual. Agencies required to have a standard treatment as usual that minimally met the same expectations at BSFT Typically services include individual, group, and family therapy sessions as well as case management
- Total: Total of all reporting groups
Arm/Group | BSFT | TAU- Treatment as Usual | Total
Number analyzed (Participants) | 245 | 235 | 480
Age, Categorical [Count of Participants; unit: Participants] — Main Study, age at baseline. A self report, demographic questionnaire was used to gather information about household composition, household income, age, race and ethnicity, gender, and age.
  Participants
    <=18 years | 245 | 235 | 480
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Categorical [Number; unit: participants in follow up study] — Follow up study, age at follow up assessment. The follow up study began 6 years after the baseline of the Main Study. All participants were over 18 at the time of the follow up study. A self report, demographic questionnaire was used to gather information about household composition, household income, age, race and ethnicity, gender, and age.
  participants in follow up study
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 140 | 121 | 261
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Main study, gender at baseline. A self report, demographic questionnaire was used to gather information about household composition, household income, age, race and ethnicity, gender, and age.
  Participants
    Female | 50 | 53 | 103
    Male | 195 | 182 | 377
Gender [Number; unit: participants in follow up study] — Follow up study, gender at follow up assessment. A self report, demographic questionnaire was used to gather information about household composition, household income, age, race and ethnicity, gender, and age.
  participants in follow up study
    Female | 26 | 27 | 53
    Male | 114 | 94 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Main study, ethnicity at baseline. A self report, demographic questionnaire was used to gather information about household composition, household income, age, race and ethnicity, gender, and age.
  Participants
    Hispanic or Latino | 107 | 106 | 213
    Not Hispanic or Latino | 133 | 125 | 258
    Unknown or Not Reported | 5 | 4 | 9
Ethnicity (NIH/OMB) [Number; unit: participants in follow up study] — Follow up study, ethnicity at follow up assessment. A self report, demographic questionnaire was used to gather information about household composition, household income, age, race and ethnicity, gender, and age.
  participants in follow up study
    Hispanic or Latino | 62 | 53 | 115
    Not Hispanic or Latino | 78 | 68 | 146
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Main Study, Adolescent Drug Use
Description: Timeline Follow Back (TLFB) measured drug use. At baseline, TLFB identified drug use in the 28-day period that preceded the baseline assessment. At all other time points the TLFB was used to collect data on daily use from the prior assessment to the current assessment. Thus, the TLFB was used to collect 365 continuous days of data on daily drug use after randomization. TLFB interview uses a calendar and other memory prompts to stimulate recall to obtain retrospective reports of daily substance use. Urine drug screens were conducted using Sure Step 10 urine drug screens and urine cups, which included temperature controlled monitoring and detection of adulterants. Urine drug screens were administered immediately prior to the administration of the TLFB to improve the chances of accurate reporting of days of use. The higher the median number, the more drug use; minimum median of drug use 0 days and maximum median of 28 days.
Time Frame: Number of self reported drug use days from 28 days prior to baseline
Population: The number of participants analyzed represents the number of participants that completed the baseline time point, assessing for the past 28 days. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use 28 days prior baseline
Groups:
- BSFT: BSFT:
  * 12-16 sessions, ranging from 8 to 24 as full dose
  * Sessions include adolescents and family members
- TAU- Treatment as Usual: TAU: Treat As Usual
  * Agencies required to have a standard treatment as usual that minimally met the same expectations at BSFT
  * Typically services include individual, group, and family therapy sessions as well as case management
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 245 | 234
days of drug use 28 days prior baseline | 3 [1 to 11] | 3 [0 to 9]
Statistical Analysis 1: Comparison: BSFT vs TAU- Treatment as Usual; Null Hypothesis: BSFT will be significantly more effective than TAU in reducing adolescent drug abuse, defined as the percentage of drug use days in 28-day periods. The outcome variable is the percentage of days of drug use within a 28-day period. This variable constructed from the Timeline-Follow-back instrument and measured as the sum of the number of days with positive use in 28-day increments. Hypothesis tested using hierarchical linear models; Test type: Superiority or Other; p = .27, Mixed Models Analysis; slope of linear trajectory of drug use = .05, 95% CI 2-sided [-.04 to .14] — The parameter estimated is the regression coefficient on the interaction of the BSFT treatment assignment and the linear time trend

2. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 1-28
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 1-28. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 1-28
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 219 | 201
days of drug use from day 1-28 | 1 [0 to 6] | 2 [0 to 8]

3. Secondary Outcome: Main Study, Externalizing Behaviors at Baseline
Description: For the Main study, an equally weighted composite of the following standardized scales was used to assess externalizing behaviors: 'Total Delinquency' from the National Youth Survey; 'Oppositional Defiant Disorder' and 'Conduct Problems' from the Diagnostic Interview Schedule for Children-Predictive Scales, 'Externalizing Scale' from the Youth Self-Report. This composite was then transformed to a z-score using the mean and standard deviation of the baseline in the entire sample. Adolescent externalizing behaviors were assessed at 4-, 8-, and 12-months post randomization.This hypothesis analyzed using hierarchical linear models. Scores ranged from -1.6 to 3.0. The higher the score, the more externalizing behavior.
Time Frame: Baseline
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing externalizing behaviors at baseline. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 245 | 235
units on a scale | -.004 (1.01) | .004 (1.03)
Statistical Analysis 1: Comparison: BSFT vs TAU- Treatment as Usual; Null hypothesis: It is hypothesized that BSFT will be significantly more effective than TAU in decreasing adolescent externalizing problem behaviors; Test type: Superiority or Other; p = .26, Mixed Models Analysis; Slope = -0.10, 95% CI 2-sided [-0.28 to 0.08] — The parameter estimated is the regression coefficient on the interaction of BSFT treatment assignment and the linear time trend

4. Secondary Outcome: Main Study, Externalizing Behavior at 4 Months Post Randomization
Description: For the Main study, an equally weighted composite of the following standardized scales was used to assess externalizing behaviors: 'Total Delinquency' from the National Youth Survey; 'Oppositional Defiant Disorder' and 'Conduct Problems' from the Diagnostic Interview Schedule for Children-Predictive Scales, 'Externalizing Scale' from the Youth Self-Report. This composite was then transformed to a z-score using the mean and standard deviation of the baseline in the entire sample. Adolescent externalizing behaviors were assessed at 4-, 8-, and 12-months post randomization.This hypothesis analyzed using hierarchical linear models. Scores ranged from -1.6 to 3.8. The higher the score, the more externalizing behavior.
Time Frame: 4 months post randomization
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for externalizing behavior at 4 months post randomization. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 191 | 185
units on a scale | -.36 (.89) | -.21 (1.07)

5. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days in days 29-56
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 29-56. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use in days 29-56
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 211 | 192
days of drug use in days 29-56 | 2 [0 to 7] | 1 [0 to 8.5]

6. Secondary Outcome: Main Study, Externalizing Behavior at 8 Months Post Randomization
Description: For the Main study, an equally weighted composite of the following standardized scales was used to assess externalizing behaviors: 'Total Delinquency' from the National Youth Survey; 'Oppositional Defiant Disorder' and 'Conduct Problems' from the Diagnostic Interview Schedule for Children-Predictive Scales, 'Externalizing Scale' from the Youth Self-Report. This composite was then transformed to a z-score using the mean and standard deviation of the baseline in the entire sample. Adolescent externalizing behaviors were assessed at 4-, 8-, and 12-months post randomization.This hypothesis analyzed using hierarchical linear models. Scores ranged from -1.6 to 3.5. The higher the score, the more externalizing behavior.
Time Frame: 8 months post randomization
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for externalizing behavior at 8 months post randomization. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 168 | 162
units on a scale | -.45 (.81) | -.39 (.99)

7. Secondary Outcome: Main Study, Externalizing Behavior at 12 Months Post Randomization
Description: For the Main study, an equally weighted composite of the following standardized scales was used to assess externalizing behaviors: 'Total Delinquency' from the National Youth Survey; 'Oppositional Defiant Disorder' and 'Conduct Problems' from the Diagnostic Interview Schedule for Children-Predictive Scales, 'Externalizing Scale' from the Youth Self-Report. This composite was then transformed to a z-score using the mean and standard deviation of the baseline in the entire sample. Adolescent externalizing behaviors were assessed at 4-, 8-, and 12-months post randomization.This hypothesis analyzed using hierarchical linear models. Scores ranged from -1.6 to 3.4. The higher the score, the more externalizing behavior.
Time Frame: 12 months post randomization
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for externalizing behavior at 12 months post randomization. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 164 | 153
units on a scale | -.45 (.93) | -.52 (.87)

8. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 57-84
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 57-84. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 57-84
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 208 | 185
days of drug use from day 57-84 | 1 [0 to 6.5] | 1 [0 to 7]

9. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 85-112
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 85-112. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 85-112
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 194 | 179
days of drug use from day 85-112 | 1 [0 to 7] | 2 [0 to 7]

10. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 113-140
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 113-140. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from days 113-140
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 186 | 176
days of drug use from days 113-140 | 1 [0 to 6] | 1 [0 to 6]

11. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 141 - 168
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 141-168. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 141-168
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 187 | 170
days of drug use from day 141-168 | 1 [0 to 8] | 1.5 [0 to 8]

12. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 169-196
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 169-196. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 169-196
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 173 | 162
days of drug use from day 169-196 | 1 [0 to 7] | 1 [0 to 9]

13. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 197-224
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 197-224. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 197-224
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 173 | 162
days of drug use from day 197-224 | 1 [0 to 10] | 1 [0 to 8]

14. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 225-252
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 225-252. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 225-252
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 165 | 161
days of drug use from day 225-252 | 2 [0 to 9] | 2 [0 to 8]

15. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 253-280
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 253-280. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 253-280
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 170 | 155
days of drug use from day 253-280 | 2 [0 to 8] | 2 [0 to 8]

16. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use from days 281-308
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 281-308. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 281-308
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 169 | 153
days of drug use from day 281-308 | 2 [0 to 10] | 2 [0 to 10]

17. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 309-336
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 309-336. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 309-336
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 162 | 149
days of drug use from day 309-336 | 2 [0 to 10] | 3 [0 to 10]

18. Primary Outcome: Main Study, Adolescent Drug Use
Description: as for outcome 1
Time Frame: Number of self reported drug use days from day 337-364
Population: The number of participants analyzed represents the number of participants that completed this time point, assessing for drug use from day 337-364. It was not necessary for the participant to complete other time points in order to be analyzed for the current time point.
Measure: Median (Inter-Quartile Range); unit: days of drug use from day 337-364
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 157 | 140
days of drug use from day 337-364 | 2 [0 to 9] | 3.5 [0 to 11]

19. Primary Outcome: Follow Up Study, Drug Use
Description: Timeline Follow Back (TLFB) measured drug use. For the Follow Up Study, the TLFB was used to identify drug use in the 90 day period that preceded the assessment. TLFB interview uses a calendar and other memory prompts to stimulate recall to obtain retrospective reports of daily substance use over the past 90 days. Urine drug screens were conducted using Sure Step 10 urine drug screens and urine cups, which included temperature controlled monitoring and detection of adulterants. Urine drug screens were administered immediately prior to the administration of the TLFB to improve the chances of accurate reporting of days of use.The higher the median number, the more drug use; minimum median of drug use 0 days and maximum median of 90 days.
Time Frame: Number of self reported drug use days 90 days prior assessment
Measure: Median (Inter-Quartile Range); unit: days of drug use 90 days prior assessmen
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 140 | 121
days of drug use 90 days prior assessmen | 19.5 [5 to 81] | 25 [6 to 82]
Statistical Analysis 1: Comparison: BSFT vs TAU- Treatment as Usual; Null Hypothesis: BSFT will be significantly more effective than TAU in the rates of drug use, defined as the percentage of drug use days in last 90 days. The primary hypothesis will be evaluated in terms of % of days of drug use in the last 90 days, assessed by the timeline follow-back. The general analytic approach will use generalized estimating equation (GEE) with negative binomial distribution comparing the BSFT and TAU participants; Test type: Superiority or Other; p = .21, GEE; Rate Ratio = .94, 95% CI 2-sided [.82 to 1.09]

20. Primary Outcome: Follow Up Study, Drug Use
Description: as for outcome 19
Time Frame: Number of self reported drug use days 90 days prior to assessment
Measure: Median (Inter-Quartile Range); unit: days of drug use 90 days prior assessmen
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 140 | 121
days of drug use 90 days prior assessmen | 8 [2 to 28] | 10 [2 to 28]

21. Secondary Outcome: Follow Up Study, Externalizing Behavior
Description: For the follow up study, externalizing behavior for the 90 days prior to the follow up was assessed using the externalizing composite of the Adult Self Report (ASR). The ASR is a 123 item self report scale designed for 18 to 59 year-old to describe their own functioning. Items are on a 3 point likert type scale (0= not true, 1=somewhat true, 2=very true or often true). The externalizing scale is comprised by the aggressive, rule braking and intrusive syndromes. The problem syndromes have been normed by sex and age (18 to 35, or 36 to 59), using a nationally representative sample. Scores were square-root transformed to more closely approximate a normal distribution. Scores ranged from 0 to 7.2. The higher the score, the more externalizing behavior. Participants were also asked to self report arrests in the past year . Externalizing was analyzed using regression
Time Frame: 90 days prior to assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 140 | 121
units on a scale | 3.1 (1.5) | 3.5 (1.5)
Statistical Analysis 1: Comparison: BSFT vs TAU- Treatment as Usual; Null hypothesis: It is hypothesized that BSFT will be significantly more effective than TAU in the level of externalizing problem behaviors; Test type: Superiority or Other; p < .006, GEE; Mean Difference (Final Values) = -.42, 95% CI 2-sided [-.71 to -.12]

22. Secondary Outcome: Main Study, Level of Family Functioning at Baseline
Description: The four components of the 'Parenting Practices Inventory' used to create a composite for use in this analysis. The four component scales from the Parenting Practices Inventory are 'Positive Parenting', 'Discipline Effectiveness,' 'Avoidance of Discipline' and 'Monitoring' scales from the Pittsburgh Youth Survey. the family functioning composite was standardized by the full sample standard deviation at baseline. Scores ranged from -3.0 to 1.8. The higher the score, the better outcome of family functioning.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 245 | 235
units on a scale | -0.03 (1.01) | 0.04 (0.99)
Statistical Analysis 1: Comparison: BSFT vs TAU- Treatment as Usual; Null hypothesis: BSFT will be significantly more effective than TAU in improving family functioning.The four components of the 'Parenting Practices Inventory' will be used to create a composite for use in this analysis. The four component scales from the Parenting Practices Inventory are 'Positive Parenting', 'Discipline Effectiveness,' 'Avoidance of Discipline' and 'Monitoring' scales from the Pittsburgh Youth Survey. Hypothesis will be analyzed as using hierarchical linear models; Test type: Superiority or Other; p = .015, Mixed Models Analysis; Slope = .12, 95% CI 2-sided [.03 to .22]

23. Secondary Outcome: Main Study, Level of Family Functioning at 4 Months Post Randomization
Description: The four components of the 'Parenting Practices Inventory' used to create a composite for use in this analysis. The four component scales from the Parenting Practices Inventory are 'Positive Parenting', 'Discipline Effectiveness,' 'Avoidance of Discipline' and 'Monitoring' scales from the Pittsburgh Youth Survey. the family functioning composite was standardized by the full sample standard deviation at baseline. Scores ranged from -2.9 to 1.8. The higher the score, the better outcome of family functioning.
Time Frame: 4 months post randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 194 | 188
units on a scale | 0.15 (1.02) | 0.21 (0.94)

24. Secondary Outcome: Main Study, Level of Family Functioning at 8 Months Post Randomization
Description: The four components of the 'Parenting Practices Inventory' used to create a composite for use in this analysis. The four component scales from the Parenting Practices Inventory are 'Positive Parenting', 'Discipline Effectiveness,' 'Avoidance of Discipline' and 'Monitoring' scales from the Pittsburgh Youth Survey. the family functioning composite was standardized by the full sample standard deviation at baseline.Scores ranged from -2.8 to 2.0. The higher the score, the better outcome of family functioning.
Time Frame: 8 months post randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 169 | 164
units on a scale | 0.31 (0.96) | 0.25 (0.97)

25. Secondary Outcome: Main Study, Level of Family Functioning at 12 Months Post Randomization
Description: The four components of the 'Parenting Practices Inventory' used to create a composite for use in this analysis. The four component scales from the Parenting Practices Inventory are 'Positive Parenting', 'Discipline Effectiveness,' 'Avoidance of Discipline' and 'Monitoring' scales from the Pittsburgh Youth Survey. the family functioning composite was standardized by the full sample standard deviation at baseline.Scores ranged from -2.6 to 2.0. The higher the score, the better outcome of family functioning.
Time Frame: 12 months post randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 169 | 158
units on a scale | 0.35 (0.96) | 0.14 (0.99)

26. Secondary Outcome: Follow Up Study, Level of Family Functioning
Description: For the follow up study, family functioning was measured by a composite of the Cohesion and Conflict scales of the Family Environment Scale. Scores ranged from 1.0 to 18.0. The higher the value, the better the level of family functioning outcome.
Time Frame: 90 days prior assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 141 | 121
units on a scale | 13.2 (4.2) | 12.4 (4.0)
Statistical Analysis 1: Comparison: BSFT vs TAU- Treatment as Usual; Test type: Superiority or Other; p = .12, GEE; Mean Difference (Net) = .68, 95% CI 2-sided [-.18 to 1.54]

27. Secondary Outcome: Main Study, Risky Sexual Behaviors at Baseline
Description: For the Main Study, the total score of the 'HIV/Sex Risk Behaviors' measure was used as the outcome. Scores ranged from -0.5 to 8.7. The higher the score, the more risky sexual behavior.
Time Frame: Baseline
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 245 | 235
units on a scale | .95 (.14) | 1.00 (.12)
Statistical Analysis 1: Comparison: BSFT vs TAU- Treatment as Usual; Null hypothesis: BSFT will be significantly more effective than TAU in decreasing sexually risky behaviors. The total score of the 'HIV/Sex Risk Behaviors' measure will be used as the outcome.Hypothesis analyzed using the hierarchical linear model; Test type: Superiority or Other; p = .12, GEE; Slope = .33, 95% CI 2-sided [-.09 to .76] — [estimate comment as in outcome 3, analysis 1]

28. Secondary Outcome: Main Study, Risky Sexual Behaviors at 4 Months Post Randomization
Description: For the Main Study, the total score of the 'HIV/Sex Risk Behaviors' measure was used as the outcome. Scores ranged from -0.5 to 10.4. The higher the score, the more risky sexual behavior.
Time Frame: 4 months post randomization
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 191 | 185
units on a scale | .89 (.12) | 1.18 (.12)

29. Secondary Outcome: Main Study, Risky Sexual Behaviors at 8 Months Post Randomization
Description: For the Main Study, the total score of the 'HIV/Sex Risk Behaviors' measure was used as the outcome. Scores ranged from -0.5 to 6.8. The higher the score, the more risky sexual behavior.
Time Frame: 8 months post randomization
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 168 | 163
units on a scale | 1.01 (.12) | 1.32 (.12)

30. Secondary Outcome: Main Study, Risky Sexual Behaviors at 12 Months Post Randomization
Description: For the Main Study, the total score of the 'HIV/Sex Risk Behaviors' measure was used as the outcome. Scores ranged from -0.5 to 6.7. The higher the score, the more risky sexual behavior.
Time Frame: 12 months post randomization
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 164 | 154
units on a scale | 1.30 (.14) | 1.44 (.12)

31. Secondary Outcome: Follow Up Study, Risky Sexual Behaviors
Description: For the Follow Up Study, sexual risk behavior was measured by examining the number of unprotected sexual acts and the number of partners and number of sex acts that included substance use the in the 90 day period that preceded the assessment; a latent factor using structural equation modeling will be used created from the Behavioral Risk Assessment. Scores ranged from -0.5 to 11.7. The higher the score, the more risky sexual behavior.
Time Frame: 90 days prior assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BSFT | TAU- Treatment as Usual
Number analyzed (Participants) | 140 | 121
units on a scale | 2.06 (.06) | 2.20 (.10)
Statistical Analysis 1: Comparison: BSFT vs TAU- Treatment as Usual; Test type: Superiority or Other; p = .23, GEE; Mean Difference (Net) = .14, 95% CI 2-sided [-.09 to .37]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Main Study:Adverse Events (AE) tracked- arrest, school suspension/drop out, runaway, kicked out of home, violence. Serious Adverse Events (SAE) tracked-physical/sexual abuse, suicidal/homicidal behavior, hospitalization, death. Follow Up Study:AE/SAE's not tracked given brief time of involvement in the study/minimal risk in completing assessment.
Groups:
- BSFT: Brief Strategic Family Therapy For Adolescent Drug Abusers: BSFT is a family therapy approach that consists of 12 to 16 sessions (each 1 to 1.5 hours long) over a 4-month period, and up to 8 "booster" sessions. Interventions are delivered to adolescents and relevant family members in non-restrictive community settings (e.g., clinics, homes, school).
- Treatment as Usual: Treatment as Usual: TAU varies depending on site, however each will offer services that include at least 1 therapy session per week (individual or group therapy) as well as participation in ancillary services (e.g., case management, self help groups, etc.) over a four month period.
Arm/Group | BSFT | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 16/245 | 16/235
Other Adverse Events (participants affected / at risk) | 144/245 | 133/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BSFT (N=245) | Treatment as Usual (N=235)
Physical/ Sexual Abuse (Social circumstances) | 2 | 2
Suicidal Behavior (Social circumstances) | 8 | 5
Homicidal Behavior (Social circumstances) | 3 | 4
Hospitalization (Social circumstances) | 8 | 8
Death (Social circumstances) | 0 | 1
Other Unexpected SAE (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BSFT (N=245) | Treatment as Usual (N=235)
Arrest (Social circumstances) | 85 | 79
Runaway (Social circumstances) | 34 | 45
Kicked out of home (Social circumstances) | 6 | 4
School suspension (Social circumstances) | 72 | 71
Violence (Social circumstances) | 31 | 23
Other Unexpected Adverse Event (Social circumstances) | 12 | 3

LIMITATIONS AND CAVEATS:
Main Study: Low rates self-reported drug use leading to only examination of prevention of relapse/escalation of drug use Follow Up Study: Variability between the time of participation in main and follow up, so no direct casuality could be concluded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No